CLINICAL TRIAL: NCT02766894
Title: Adequate Depth of Anesthesia: the Anesthesiologist's Assessment and the EEG Processed Monitoring
Status: Completed | Type: Observational
Sponsor: Kepler University Hospital (Other)
Responsible Party: Principal Investigator, Wolfgang Puchner MD, MD, Kepler University Hospital
Other Study IDs: C-109-16
Record Dates: First submitted 2016-05-01; First posted 2016-05-10 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: EEG monitoring — EEG will be performed. Data obtained will be analyzed using software. Anesthesiologists will enter their assumption in a blinded fashion and data obtained will be compared with EEG data

SUMMARY:
Comparison of conventional assessment of anesthetic depth by anesthesiologists (moderate, deep or light anesthesia) with EEG monitoring (Narcotrend® state/index). In case of mismatch statistical analysis for underlying factors are done.

DETAILED DESCRIPTION:
In this observational study estimation of anesthetic depth by anesthesiologists is compared with the EEG based monitoring Narcotrend®. 10-20 voluntary anesthesiologists of the Kepler University Hospital, unfamiliar with EEG-monitoring during anesthesia, assess depth of anesthesia (moderate, deep or light level) during a steady-state period by clinical signs and measured or calculated concentrations of anesthetics. Concurrently Narcotrend® provides data of anesthetic depth (index, stadium) blinded for the anesthesiologist. Each anesthesiologist is included 30 times during study period. The aim of this study is to define conformity between subjective and objective assessment of narcotic depth. In the cases of divergence data of the patient (age, body mass index, comorbidity…), data of the anesthesiologist (age, years of practice…), data of anesthesia (balanced anesthesia, target controlled infusion, endtidal concentration of volatile anesthetic…) and data of the operation (eye surgery, cardiac surgery…) will be analyzed by statistics with regard to underlying or concomitant factors. These findings could help to develop recommendations in the use of EEG-processed monitoring to improve subjective assessment and facilitate an adequate depth of anesthesia to be provided for every patient.

ELIGIBILITY:
Inclusion Criteria:

* operation under general anesthesia
* duration of surgery ≥ 10 minutes
* informed consent
* ASA physical status 1-4
* age 1-110y
* performance check of Narcotrend

Exclusion Criteria:

* proximity of EEG electrodes to the operating field
* frontal skin lesion
* frontal cerebral pathology
* hypoxic brain damage
* hypothermia (≤33°C)
* language barrier

Ages: 1 Year to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients:
  Randomization of patients (m/w) after informed consent. For detailed inclusion criteria see corresponding section.
  Patients are randomly assigned to anesthesiologist. Anesthesiologists are blinded and must assume anesthesia level. Evaluation will be performed by study leader.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2016-05; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Comparison of subjective (anesthesiologist) vs. objective (Narcotrend) assessment of anesthesia depth. | up to 1 year
  Depth of anesthesia will be assessed by the anesthesiologist in an subjective way. During a defined period of stable anesthesia state, the indicated subjective depth levels will be assessed by the anesthesiologist and will be compared to those obtained by narcotrend (Narcotrend-Index). Anesthesiologists will assess by deep, moderate and superficial depth of anesthesia. Narcotrend indices will also be assigned to three groups (superficial, moderate, deep levels). After the procedure, both systems will be compared. In the case of non-correlation, other factors like i.e. patient's age, comorbidities, years of practice of the anesthesiologist etc. will be analysed for any other type of correlation.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Meier, MD, PhD, Study Chair — Kepler UH, Dept. of Anesthesiology

IPD SHARING:
Plan to Share IPD: Yes
Data will be accessible on central server to observers after completion of the study

REFERENCES:
- [Background] Kreuer S, Bruhn J, Stracke C, Aniset L, Silomon M, Larsen R, Wilhelm W. Narcotrend or bispectral index monitoring during desflurane-remifentanil anesthesia: a comparison with a standard practice protocol. Anesth Analg. 2005 Aug;101(2):427-434. doi: 10.1213/01.ANE.0000157565.00359.E2. PMID 16037157
- [Background] Bauerle K, Greim CA, Schroth M, Geisselbrecht M, Kobler A, Roewer N. Prediction of depth of sedation and anaesthesia by the Narcotrend EEG monitor. Br J Anaesth. 2004 Jun;92(6):841-5. doi: 10.1093/bja/aeh142. Epub 2004 Apr 2. PMID 15064250
- [Derived] Puchner WF, Dunser MW, Paulus P, Neuner MP, Mayer CL, Pomberger IM, Hackl R, Meier JM. A comparative study on adequate anesthesia depth: clinical judgement and the Narcotrend(R) measurement. Can J Anaesth. 2020 Jun;67(6):664-673. doi: 10.1007/s12630-020-01602-x. Epub 2020 Mar 3. PMID 32128723